CLINICAL TRIAL: NCT03619239
Title: A Phase 1b, Dose-escalation Study to Evaluate the Safety, Tolerability, and the Lymphocyte Increasing Effects of GX-I7 Intramuscular Administration in Patients With Glioblastoma
Brief Title: Dose-escalation Study to Evaluate the Safety and Tolerability of GX-I7 in Patients With Glioblastoma
Acronym: GBM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GX-I7-CA-004
Record Dates: First submitted 2018-06-26; First posted 2018-08-07 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-03

CONDITIONS: Newly Diagnosed Glioblastoma
Keywords: Phase 1b
MeSH Terms: interventions — efineptakin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Patients will receive treatment with GX-I7 at a pre-determined dose (Level I) on Day1 of each cycle.
  Interventions: Drug: GX-I7
- Cohort 2 (Experimental): Patients will receive treatment with GX-I7 at a pre-determined dose (Level II) on Day1 of each cycle.
  Interventions: Drug: GX-I7
- Cohort 3 (Experimental): Patients will receive treatment with GX-I7 at a pre-determined dose (Level III) on Day1 of each cycle.
  Interventions: Drug: GX-I7
- Cohort 4 (Experimental): Patients will receive treatment with GX-I7 at a pre-determined dose (Level IV) on Day1 of each cycle.
  Interventions: Drug: GX-I7
- Cohort 5(Dose-expansion) (Experimental): Optimal fixed dose of GX-I7 from Dose-escalation stage on Day1 of each cycle (Maximum tolerable dose or Maximum efficacious dose or Maximum administered dose level or consecutive lower or upper dose level which does not exceed Maximum tolerable dose based on Safety Monitoring Committee(SMC) decision)
  Interventions: Drug: GX-I7

INTERVENTIONS:
Drug: GX-I7 — During Treatment Period, patients will receive the assigned dose of GX-I7 intramuscular injection every 4~12 weeks per cycle up to 6 cycles in the absence of unacceptable toxicity or clinically compelling evidence of disease progression.

SUMMARY:
Patients will be enrolled in two stages:

* Dose-escalation stage: Approximately 12-24 patients will be enrolled.

DETAILED DESCRIPTION:
Detailed Description:

• Dose-escalation stage : designed as classical 3+3 to determine MTD(Maximum tolerable dose), RP2D(Recommended Phase 2 Dose) and DLT(Dose-limiting toxicity)s to evaluate approximately four dose levels of GX-I7

* pre-determined dose(Level I)~ pre-determined dose(Level IV)

ELIGIBILITY:
[Inclusion Criteria]

1. Ability to understand and willingness to sign a written informed consent document (ICF).
2. Age ≥ 19 years
3. Able to comply with the study protocol, in the investigator's judgment
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

[Exclusion Criteria] General Exclusion Criteria

1. Unable to comply with study and follow-up procedures
2. Is pregnant or breastfeeding
3. Have clinically significant cardiac disease (New York Heart Association, Class II or greater) including myocardial infarction, unstable arrhythmias, and/or unstable angina in the past 3 months
4. Have clinically significant liver disease, including alcoholic, or other hepatitis, cirrhosis, and inherited liver disease or current alcohol abuse

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
DLT(Dose-Limiting Toxicity) Assessment | Through study completion, an average of 2 years
  Incidence and nature of DLT(Dose-Limiting Toxicity)s
Incidence, nature and severity of Adverse events | Through study completion, an average of 2 years
  Incidence, nature and severity of adverse events graded according to NCI CTCAE v4.0

SECONDARY OUTCOMES:
PD(pharmacodynamic) profile [ALC result] | Through study completion, an average of 2 years
  Changes of ALC(Absolute lymphocyte count) from the baseline
Anti-tumor Activity [OS] | Through study completion, an average of 2 years
  Objective response(OS) defined as the time from the date of diagnosis to the death from any cause
Anti-tumor Activity [PFS] | Through study completion, an average of 2 years
  Progression-free survival (PFS) defined according to iRANO(Immunotherapy Response Assessment for Neuro-Oncology)
Immunogenicity[ ADA and neutralizing antibody] | Through study completion, an average of 2 years
  Incidence of anti-GX-I7 antibody (ADA) and neutralizing antibody during the study
Exploratory Biomarker [serum Interleukin-7] | Through study completion, an average of 2 years
  Changes in serum Interleukin-7

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Seoul St. Mary's Hospital, Seoul, Seocho, South Korea